CLINICAL TRIAL: NCT00694616
Title: Prevalence of Metabolic Syndrome in Obstructive Sleep Apnea and the Effect of Treatment With Auto-titrating Continuous Positive Airway Pressure (Auto-CPAP) on Metabolic Syndrome
Brief Title: Prevalence of Metabolic Syndrome in Obstructive Sleep Apnea (OSA) and Effect of Treatment With Continuous Positive Airway Pressure (Auto-CPAP) on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, S.K.SHARMA, Professor and Head, All India Institute of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SKS/OSA/CPAP/2008
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Obstructive Sleep Apnea; Metabolic Syndrome
Keywords: Obstructive sleep apnea; Metabolic syndrome; Insulin resistance; Hypertension; Dyslipidemia; Continuous positive airway pressure (CPAP)
MeSH Terms: conditions — Sleep Apnea, Obstructive; Metabolic Syndrome; Insulin Resistance; Hypertension; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): 3 months of therapeutic CPAP (auto-titrating CPAP) followed by 3 months of non-therapeutic sham-CPAP with 1 month of wash-out in between
  Interventions: Device: AutoSet Spirit
- 2 (Other): 3 months of non-therapeutic sham-CPAP followed by 3 months of therapeutic CPAP (auto-titrating CPAP) with 1 month of wash-out in between
  Interventions: Device: Modified-AutoSet Spirit

INTERVENTIONS:
Device: AutoSet Spirit — 3 months of therapeutic CPAP (auto-titrating CPAP) followed by 3 months of non-therapeutic sham-CPAP with 1 month of wash-out in between
  Other Names: AutoSet Spirit(TM), ResMed India Ltd.
  Arms: 1
Device: Modified-AutoSet Spirit — 3 months of non-therapeutic sham-CPAP followed by 3 months of therapeutic CPAP (auto-titrating CPAP) with 1 month of wash-out in between
  Other Names: Modified-AutoSet Spirit(TM), ResMed India Ltd.
  Arms: 2

SUMMARY:
Metabolic syndrome is a constellation of risk factors for cardiovascular disease. The prevalence of metabolic syndrome in persons with obstructive sleep apnea syndrome (OSAS) is known to be very high, about 70%. However, it is unclear whether this association is causal or not. Results of earlier studies have been conflicting. The investigators hypothesize that treatment with auto-titrating continuous positive airway pressure (auto-CPAP) for a duration of 3 months improves the metabolic syndrome in subjects with OSAS.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a condition in which there is collapse of the upper airway during sleep, as a result of which there is a decrease or complete cessation of airflow. This leads to repeated episodes of hypoxia during sleep and sleep fragmentation. OSA is a highly prevalent though under-recognized clinical problem. The Wisconsin study estimated a prevalence of 24% in males and 9% in females. A population-based study in Delhi, India found the prevalence of OSA to be 13.7% and that of obstructive sleep apnea syndrome (OSAS) to be 3.8%.

OSA is associated with various systemic complications such as neurocognitive dysfunction, cardiovascular disease, insulin resistance, and dyslipidemia. There is an increased risk of motor vehicle and occupational accidents in people suffering from OSAS.

Metabolic syndrome is the co-occurrence of several cardiovascular risk factors such as abdominal obesity, hypertension, impaired glucose tolerance and dyslipidemia. Presence of OSA together with metabolic syndrome is known as 'Syndrome Z'. Although many studies have shown that OSA is associated with metabolic syndrome, the exact causal relationship between these two entities is not proven.

Continuous positive airway pressure (CPAP) is the standard treatment for OSA with significant symptoms. However, it is a costly treatment option, and poor compliance is an important limiting factor. CPAP treatment has been shown to improve the daytime somnolence and neurocognitive function in people with OSAS. However, its effect on metabolic syndrome in people with OSAS is unclear.

This study aims to assess the effect of CPAP treatment on metabolic syndrome in patients with OSAS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderately severe OSAS (AHI >= 15 with excessive daytime sleepiness) also having metabolic syndrome, and have never received treatment for OSAS, diabetes mellitus and hypertension

Exclusion Criteria:

* Diabetic subjects will be excluded if any one of the following is present

  1. Proliferative diabetic retinopathy
  2. Nephropathy (serum creatinine >1.8 mg/dL)
  3. Clinically manifest neuropathy defined as absent ankle jerks.
  4. Severe hyperglycemia (FBS >200 mg/dL)
* Hypertensive subjects will be excluded if any one of the following is present

  1. Symptomatic coronary artery disease
  2. Symptomatic peripheral vascular disease
  3. Past history of cerebrovascular accident
  4. Known case of aortic aneurysm or left ventricular dysfunction
  5. Nephropathy (serum creatinine >1.8 mg/dL)
  6. Marked elevation in blood pressure (BP >180/110 mm Hg on two occasions)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects satisfying the National Cholesterol Education Program-Adult Treatment Panel (NCEP-ATP III) criteria for the diagnosis of metabolic syndrome | 3 months

SECONDARY OUTCOMES:
Individual components of the NCEP-ATP III criteria (FBS, BP, LDL cholesterol, HDL cholesterol, triglycerides) and insulin resistance (assessed by HOMA-IR) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, M.D., Ph.D., Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, New Delhi, India

REFERENCES:
- [Derived] Sharma SK, Agrawal S, Damodaran D, Sreenivas V, Kadhiravan T, Lakshmy R, Jagia P, Kumar A. CPAP for the metabolic syndrome in patients with obstructive sleep apnea. N Engl J Med. 2011 Dec 15;365(24):2277-86. doi: 10.1056/NEJMoa1103944. PMID 22168642 (Retraction: PMID 24171540 Sharma SK, Agrawal S, Damodaran D, Sreenivas V, Kadhiravan T, Lakshmy R, Jagia P, Kumar A. N Engl J Med. 2013 Oct 31;369(18):1770)